CLINICAL TRIAL: NCT06879925
Title: The Effects of Qi-gong on Physiology and Quality of Life in Patients with Post-acute Sequelae of Covid-19
Brief Title: Physiological and QoL Benefits of Qi-Gong in Post-acute Sequelae of Covid-19
Acronym: QG-PASC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: POCHIWU (Other)
Responsible Party: Sponsor-Investigator, POCHIWU, nurse、master's candidate, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CTH-113-3-5-030; NTUNHS (Registry Identifier: National Taipei University of Nursing and Health Sciences)
Record Dates: First submitted 2025-02-15; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: PASC Post Acute Sequelae of COVID 19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: Experimental Group:QIGONG Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qi-Gong Group (Experimental): Experimental Group :Qi-Gong(yijinjing)
  Interventions: Behavioral: QI-GONG and control
- routine care Group (No Intervention): Control Group:routine care

INTERVENTIONS:
Behavioral: QI-GONG and control — QIGONG
  Arms: Qi-Gong Group

SUMMARY:
The goal of this clinical trial is to determine whether Qi-Gong can improve physiological function and quality of life (QoL) in individuals with post-acute sequelae of SARS-CoV-2 infection (PASC).

Study Objectives:

To assess whether Qi-Gong improves physiological function in individuals with PASC.

To evaluate whether Qi-Gong enhances quality of life in individuals with PASC.

Study Design:

If a comparison group is included, researchers will compare Qi-Gong with standard care to assess its effectiveness.

Participant Involvement:

Practice Qi-Gong three times per week for three months. Record physiological data monthly.

ELIGIBILITY:
Inclusion Criteria:

* PASC
* above 20 y/o

Exclusion Criteria:

* Those who cannot cooperate
* Severe schizophrenia

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test (Forced vital capacity) | From enrollment to the end of treatment at 12 weeks
  FVC，over 80% is better
Pulmonary Function Test (FEV1) | From enrollment to the end of treatment at 12 weeks
  FEV1，over 80% is better
Pulmonary Function Test (FVCFEV1) | From enrollment to the end of treatment at 12 weeks
  FVCFEV1，over 80% is better
Heart rate variability | From enrollment to the end of treatment at 12 weeks
  Low Frequency,40%-60%
Heart rate variability | From enrollment to the end of treatment at 12 weeks
  High Frequency,40%-60%
Heart rate variability | From enrollment to the end of treatment at 12 weeks
  LF/HF,0.6-2.5
Heart rate variability | From enrollment to the end of treatment at 12 weeks
  Heart rate variability ,25ms-70ms
Quality of Life(The short version of the World Health Organization Quality of Life ，WHOQOL-BREF) | From enrollment to the end of treatment at 12 weeks
  WHOQOL-BREF 4 domains,and each one score is 4 - 20. more score more better

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hua Wang, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (2):
- Taiwan (2):
  - Renhe nursing home, New Taipei City
  - Fuxi nursing home, Taipei

IPD SHARING:
Plan to Share IPD: No